CLINICAL TRIAL: NCT02476773
Title: Phase 1 Study of the Safety and Immunogenicity of Na-APR-1 (M74)/Alhydrogel® Co-administered With Na-GST-1/Alhydrogel® in Brazilian Adults
Brief Title: Study of Na-APR-1 (M74)/Alhydrogel® Co-administered With Na-GST-1/Alhydrogel in Brazilian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Centro de Pesquisas René Rachou (Other Government); Johns Hopkins University (Other); University of California, San Francisco (Other); George Washington University (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SVI-DBL-01
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Hookworm Vaccine; Na-APR-1 (M74)/Alhydrogel® Hookworm Vaccine; Na-GST-1/Alhydrogel® Hookworm Vaccine
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): * 5 subjects will receive 10µg Na-APR-1 (M74)/Alhydrogel with Sterile Saline Placebo administered to the alternate arm.
  * 5 subjects will receive 10µg Na-APR-1 (M74)/Alhydrogel with 100µg Na-GST-1/Alhydrogel plus GLA-AF administered to the alternate arm.
  Interventions: Biological: Na-GST-1/Alhydrogel plus GLA-AF; Biological: Na-APR-1 (M74)/Alhydrogel; Biological: Sterile Saline Placebo
- Group 2 (Experimental): * 5 subjects will receive 10µg Na-APR-1 (M74)/Alhydrogel plus GLA-AF, with Sterile Saline Placebo administered to the alternate arm.
  * 5 subjects will receive 10µg Na-APR-1 (M74)/Alhydrogel plus GLA-AF, with 100µg Na-GST-1/Alhydrogel plus GLA-AF administered to the alternate arm.
  Interventions: Biological: Na-GST-1/Alhydrogel plus GLA-AF; Biological: Na-APR-1 (M74)/Alhydrogel plus GLA-AF; Biological: Sterile Saline Placebo
- Group 3 (Experimental): * 5 subjects will receive 30µg Na-APR-1 (M74)/Alhydrogel, with Sterile Saline Placebo administered to the alternate arm.
  * 5 subjects will receive 30µg Na-APR-1 (M74)/Alhydrogel, with 100µg Na-GST-1/Alhydrogel plus GLA-AF administered to the alternate arm.
  Interventions: Biological: Na-GST-1/Alhydrogel plus GLA-AF; Biological: Na-APR-1 (M74)/Alhydrogel; Biological: Sterile Saline Placebo
- Group 4 (Experimental): * 5 subjects will receive 30µg Na-APR-1 (M74)/Alhydrogel plus GLA-AF, with Sterile Saline Placebo administered to the alternate arm.
  * 5 subjects will receive 30µg Na-APR-1 (M74)/Alhydrogel plus GLA-AF, with 100µg Na-GST-1/Alhydrogel plus GLA-AF administered to the alternate arm.
  Interventions: Biological: Na-GST-1/Alhydrogel plus GLA-AF; Biological: Na-APR-1 (M74)/Alhydrogel plus GLA-AF; Biological: Sterile Saline Placebo
- Group 5 (Experimental): * 5 subjects will receive 100µg Na-APR-1 (M74)/Alhydrogel, with Sterile Saline Placebo administered to the alternate arm.
  * 5 subjects will receive 100µg Na-APR-1 (M74)/Alhydrogel, with 100µg Na-GST-1/Alhydrogel plus GLA-AF administered to the alternate arm.
  Interventions: Biological: Na-GST-1/Alhydrogel plus GLA-AF; Biological: Na-APR-1 (M74)/Alhydrogel; Biological: Sterile Saline Placebo
- Group 6 (Experimental): * 5 subjects will receive 100µg Na-APR-1 (M74)/Alhydrogel plus GLA-AF, with Sterile Saline Placebo administered to the alternate arm.
  * 5 subjects will receive 100µg Na-APR-1 (M74)/Alhydrogel plus GLA-AF, with 100µg Na-GST-1/Alhydrogel plus GLA-AF administered to the alternate arm.
  Interventions: Biological: Na-GST-1/Alhydrogel plus GLA-AF; Biological: Na-APR-1 (M74)/Alhydrogel plus GLA-AF; Biological: Sterile Saline Placebo

INTERVENTIONS:
Biological: Na-GST-1/Alhydrogel plus GLA-AF
Biological: Na-APR-1 (M74)/Alhydrogel
  Arms: Group 1; Group 3; Group 5
Biological: Na-APR-1 (M74)/Alhydrogel plus GLA-AF
  Arms: Group 2; Group 4; Group 6
Biological: Sterile Saline Placebo

SUMMARY:
Na-GST-1 and Na-APR-1 are proteins expressed during the adult stage of the Necator americanus hookworm life cycle that are thought to play a role in the parasite's degradation of host hemoglobin for use as an energy source. Vaccination wtih recombinant GST-1 or APR-1 has protected dogs and hamsters from infection in challenge studies. This study will evaluate the safety and immunogenicity of co-administering Na-GST-1 and Na-APR-1 to healthy Brazilian adults living in an area of endemic hookworm infection.

DETAILED DESCRIPTION:
Double blind, randomized, controlled, dose-escalation Phase 1 clinical trial in hookworm exposed adults living in the area of Americaninhas, Minas Gerais, Brazil. Subjects will receive three doses of the assigned vaccine delivered intramuscularly on approximately Days 0, 56, and 112.

Safety will be measured from the time of each study vaccination (Day 0) through 14 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events.

Unsolicited non-serious adverse events (AEs) will be collected from the time of the first study vaccination through approximately 1 month after each study vaccination. New-onset chronic medical conditions and Serious Adverse Events (SAEs) will be collected from the time of the first study vaccination through approximately 9 months after the third study vaccination (final visit). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 14 days after each vaccination.

Immunogenicity testing will include IgG antibody responses to each vaccine antigen, by an indirect enzyme-linked immunosorbent assay (ELISA) and also by ImmunoCAP, on serum obtained prior to each study vaccination and at time points after each vaccination; antibody affinity by Surface Plasmon Resonance; functional activity of vaccine-induced antibodies via in vitro enzyme neutralization assays; and, antigen-specific memory B cell responses.

Recruitment and enrollment into the study will occur on an ongoing basis, with each group being recruited and vaccinated in sequence.

60 subjects will be enrolled into 6 groups of 10.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females between 18 and 45 years, inclusive.
2. Good general health as determined by means of the screening procedure.
3. Available for the duration of individual subject study participation (16 months).
4. Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

1. Pregnancy as determined by a positive urine hCG (if female).
2. Subject unwilling to use reliable contraception (as described in Section 2.3.1) from 30 days prior to the first immunization and up until one month following the third immunization (if female and not surgically sterile, abstinent or at least 2 years post-menopausal, or determined otherwise by medical evaluation to be sterile).
3. Currently lactating and breast-feeding (if female).
4. Inability to correctly answer all questions on the informed consent comprehension questionnaire.
5. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies (a history of essential hypertension that is well controlled by medication will not be considered exclusionary.)
6. Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric condition that would make compliance with study visits/procedures difficult (e.g., subject with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide).
7. Known or suspected immunodeficiency.
8. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
9. Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing with the exception of greater than trace blood detected in females during menses).
10. Laboratory evidence of hematologic disease (absolute leukocyte count <3200/mm3; absolute leukocyte count >10.8 x 103/mm3; hemoglobin <11.4 g/dl [females] or <12.1 g/dl [males]; or, platelet count <130,000/mm3).
11. Serum glucose (random) greater than 1.2-times the upper reference limit.
12. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
13. Participation in another investigational vaccine or drug trial within 30 days of starting this study.
14. Previous receipt of the Na-GST-1/Alhydrogel® hookworm vaccine.
15. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
16. History of a severe allergic reaction or anaphylaxis.
17. Severe asthma as defined by the need for daily use of inhalers or emergency clinic visit or hospitalization within the last 6 months.
18. Positive test for hepatitis B surface antigen (HBsAg).
19. Positive confirmatory test for HIV infection.
20. Positive confirmatory test for hepatitis C virus (HCV) infection.
21. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of the volunteer's expected first vaccination in this study or planned use up to one month following the last vaccination.
22. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to the volunteer's expected first vaccination in the study.
23. History of a surgical splenectomy.
24. Receipt of blood products within the past 6 months.
25. Anti-Na-GST-1 IgE antibody level above 0.35 kUA/L by the ImmunoCAP method.
26. Anti-Na-APR-1 IgE antibody level above ELISA reactivity threshold.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited injection site and systemic reactogenicity, graded by severity, on the day of each study vaccination through 14 days after each study vaccination. | 14 days post-vaccination
Frequency of study vaccine-related serious adverse events from the time of the first study vaccination through approximately 9 months after the last study vaccination. | Day 380
Frequency of clinical safety laboratory adverse events. | Day 380
Frequency of unsolicited adverse events, graded by severity, from the time of each study vaccination through approximately 1 month after each study vaccination. | 30 days post-vaccination
Frequency of new-onset chronic medical conditions through approximately 9 months after the third study vaccination. | Day 380
Frequency of Adverse Events of Special Interest through approximately 9 months after the third study vaccination. | Day 380

SECONDARY OUTCOMES:
The IgG level by an indirect enzyme-linked immunosorbent assay (ELISA) on approximately Day 126. | Day 126

OTHER OUTCOMES:
The IgG antibody response, by an indirect enzyme-linked immunosorbent assay (ELISA) at approximately 7, 14, and 28 days after each vaccination, and approximately 3, 6, and 9 months after the third dose. | 7, 14, and 28 days after each vaccination, and approximately 3, 6, and 9 months after the third dose

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, Principal Investigator — George Washington University; Rodrigo Correa-Oliveira, PhD, Study Director — Centro de Pesquisas René Rachou
Locations (1):
- Americaninhas Vaccine Center, Americaninha, Minas Gerais, Brazil

DOCUMENTS (2):
  • Study Protocol (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT02476773/Prot_000.pdf
  • Informed Consent Form (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT02476773/ICF_001.pdf